CLINICAL TRIAL: NCT02369042
Title: KYMA Device: External Measure of Thoracic Fluid and Vital Signs
Acronym: Ease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Dr. Eugene Chung, MD, The Christ Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ChristH
Record Dates: First submitted 2014-10-28; First posted 2015-02-23 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2015-02

CONDITIONS: Congestive Heart Failure(CHF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort I (Experimental): Patients admitted with the primary diagnosis of HF and are currently being assessed with clinically indicated hemodynamic monitoring.The Kyma device will be worn by the patient and data collected from the device will be compared to the data collected through hemodynamic monitoring. The device will be worn for 60 days post hospital discharge.
  Interventions: Device: Kyma Device u-Cor System
- Cohort II (Experimental): Patients admitted with the primary diagnosis of HF and are being assessed with or without hemodynamic monitoring. The Kyma device will be worn by the patient and data collected from the device will be compared to the data collected while the patient is hospitalized. The device will be worn for 60 days post hospital discharge.
  Interventions: Device: Kyma Device u-Cor System

INTERVENTIONS:
Device: Kyma Device u-Cor System — The Kyma uCor system externally measures thoracic fluid content, heart rate, respiratory rate, posture and movement. The system includes a flat antenna that is attached to the patient's torso with a bandage-like sticker. The antenna transmits radio waves and receives their reflections from the body for several seconds every few hours throughout the day.The data is recorded and collected then compared to traditional clinical parameters.

SUMMARY:
External measure of thoracic fluid content (TFC) combined with vital signs (HR,respiratory rate(RR), posture and movements) using the technology developed by Kyma Medical Technologies while tracking clinical changes in acute in-hospital and chronic outpatient heart failure patients.

DETAILED DESCRIPTION:
This is a prospective, single center, non-randomized study designed to correlate Kyma measurements and in-hospital parameters as well as the changes in TFC and vital signs with clinical changes in the outpatient setting for 60 days post-discharge. The patient and hospital study personnel will be blinded to the Kyma data captured by the device. No intervention will be performed on the patient based on the Kyma device data, this is an observational study.

The goals of the study are:

1. Follow thoracic fluid and vital signs in acute, hospitalized heart failure(HF) patients with evidence of volume overload to evaluate this combined parameter in relation to decongestion (time to clear lung auscultation or clearing of congestion on chest x-ray or decrease in BNP by 50%), clinical symptoms, physical exam, and biomarker results.
2. Evaluate the relationship between lung decongestion as externally measured and hemodynamic parameters as measured by pulmonary artery catheter in a subset of patients
3. Correlate changes in thoracic fluid content and vital signs with clinical changes in the outpatient setting for 60 days post-discharge.
4. Evaluate the feasibility of implementing a physician-directed, patient- managed model of diuretic and vasodilator adjustment.

Patients will be approached for enrollment within 24 hours of presentation to the hospital. The Kyma device will be applied to the patient. Data will be automatically collected by the device: TFC will be measured every 30 minutes and vital signs will be measured several times an hour.

Information collected at baseline by the study coordinators will include medications, lab work (CBC, Chemistry, BNP), ejection fraction(EF), weight, vital signs, and lung auscultation for both Cohorts.

Cohorts I and II may be enrolled concurrently. For patients enrolled in Cohort I, PA readings will be recorded at baseline and 3 times daily until the pulmonary artery(PA) catheter is removed.

While hospitalized, all patients will have daily weights, intake/output, Physical Exams(edema, jugular venous distention(JVP), lung exam) and vital signs will be recorded twice daily. Lab results will be recorded as well as any changes in medication.

After hospital discharge, the patients will wear the Kyma device for an additional 60 days. Patients will be contacted by telephone at 10 days, 30 days, and 60 days post-discharge for weight measurements, medication changes, and assessment of any Office Visits, or ER/Hospitalizations for SOB.

The Minnesota Living with Heart Failure Questionnaire will be administered at hospital discharge and 30 and 60 days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Cohort I

  1. Men or women over 18 years of age
  2. Admitted for primary diagnosis of HF
  3. Already assigned for indwelling PA catheter monitoring
  4. BNP > 400
  5. Two of the following: edema, JVP>7cm, rales
  6. Currently being assessed with clinically indicated hemodynamic monitoring

Cohort II

1. Men or women over 18 years of age
2. Admitted with the primary diagnosis of HF
3. BNP > 400
4. Two of the following: edema, JVP> 7cm, rales
5. Patients with or without hemodynamic monitoring in use

Exclusion Criteria:

Cohort I and II

1. Patients with allergies or skin sensitivities to electrode hydrogel and/or acrylic based adhesive
2. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03-20 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Validate the ability of externally monitored thoracic fluid content as a measure of HF. | 60 days
  Accomplished by comparing the data measured by the Kyma Device(HR, RR, thoracic fluid content) with the same clinical data collected while in the hospital.

SECONDARY OUTCOMES:
Assess the effectiveness of remote monitoring in detecting outpatient decompensation. | 60 days
  Compare the data collected by the Kyma Device (HR, RR, movement, thoracic fluid content) to any clinical changes related to HF in the outpatient setting.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Chung, MD, Principal Investigator — The Lindner Research Center at The Christ Hospital
Locations (1):
- The Lindner Research Center at The Christ Hospitak, Cincinnati, Ohio, United States